CLINICAL TRIAL: NCT06311058
Title: The Effect of Protein Supplementation on Muscle Atrophy After ACL Reconstruction
Brief Title: Protein Supplementation After ACL Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PRO00032531
Record Dates: First submitted 2024-02-16; First posted 2024-03-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: ACL Reconstruction
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Subjects are randomized to 1 of 3 intervention groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Protein Supplement Group (Experimental): Participants in this group will receive 25g of whey protein isolate twice a day for 12 weeks.
  Interventions: Dietary Supplement: Whey protein isolate
- Protein + Amino Acid Supplement Group (Experimental): * Protein drink - 25g of whey protein isolate
  * Amino Acid Blend - 7g of protein (4g Leucine, 1g iso leucine, 1g valine, 1g arginine)
  Twice a day for 12 weeks
  Interventions: Dietary Supplement: Whey protein isolate; Dietary Supplement: Protein + BAA
- Placebo Group (Placebo Comparator): • isocaloric-matched (25g) maltodextrin supplement
  Twice a day for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey protein isolate — 25g of whey protein isolate
  Arms: Protein + Amino Acid Supplement Group; Protein Supplement Group
Dietary Supplement: Protein + BAA — * Protein drink - 25g of whey protein isolate
  * Amino Acid Blend - 7g of protein (4g Leucine, 1g iso leucine, 1g valine, 1g arginine)
  Arms: Protein + Amino Acid Supplement Group
Dietary Supplement: Placebo — • isocaloric-matched (25g) maltodextrin supplement
  Arms: Placebo Group

SUMMARY:
The purpose of the study is to assess the longitudinal post-operative care effects of protein supplementation on muscle atrophy in the post-operative period following ACL reconstruction. The main outcome will be muscle size/mass as measured using dual energy x-ray absorptiometry (DEXA) scanning. The primary objective is to assess for any beneficial impact of protein supplementation, with implications of standardizing a recommended protocol for protein supplementation after ACL reconstruction.

Secondary outcomes will be to evaluate the survey data from the KOOS JR and Tampa Scale surveys, as well as functional measures recorded during physical therapy.

DETAILED DESCRIPTION:
This study is designed to evaluate non-interventional longitudinal post-operative clinical improvement. The proposed study is a randomized non-interventional, double blind study. Subjects will include patients age 16 to 40 undergoing primary ACL reconstruction for an acute ACL tear. Demographic information including age, sex, BMI, and sport participation will be obtained from patients at the time of recruitment.

Subjects will be randomized to one of three categories: 1)placebo, 2)protein supplementation, or 3)protein supplementation with amino acids. The probability is is a 1 in 3 chance to be enrolled in each group. Participants will be provided the supplement drink immediately following surgery and will be asked to consume the supplement 2-times daily following ACL reconstruction for a total of 12 weeks post-op. In addition, participants will be asked to complete a weekly food diary in which they track their diet for 2 week days and 1 weekend day each week for all 12 weeks. This will help account for dietary proteins. Subjects will also be asked to complete the KOOS Jr and Tampa Scale surveys (attached in the application) through Houston Methodist's Redcap system at each time point (Pre-op, 4, 8 and 12 weeks postop).

Briefly, BCAAs (particularly leucine) represent primary triggers for the stimulation of protein synthesis via signaling through the mammalian target of rapamycin complex 1 pathway (mTORC1) in skeletal muscle and other tissues. Whey hydrolysate is a complete protein source that is considered to be "fast absorbing." Casein is a complete protein source that is "slow absorbing" relative to whey.9 All protein sources used in this investigation are commercially available nutritional supplements. The placebo will include a crystallite drink.

Standard of care clinic assessments such as bilateral muscle strength and stability screening will be performed in all patients at 8 and 12 weeks of rehabilitation. Time to return to sport for those subjects participating in a recreational or professional sport activities will also be recorded. Lastly, quadriceps muscle mass measured through dual energy x-ray absorptiometry (DEXA) scanning. Participants in all 3 groups will undergo DEXA scanning at once pre-operatively, 4 weeks post-op,8 weeks, post-op and 12 weeks post-op following ACL reconstruction.

The Tampa Scale and KOOS JR surveys will be administered at each study visit. The purpose of these surveys are to evaluate patient perception of surgery and their injury. As stated in the purpose, these will act as secondary outcomes to this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include patients age 16 to 40 undergoing primary ACL reconstruction for an acute ACL tear with the PI or Sub-investigators

Exclusion Criteria:

* Subjects will not be included if they meet one of the following criteria

  * History of meniscectomy or meniscus repair
  * Obesity (BMI>35)
  * Diabetes
  * Cardiovascular, renal, liver or pulmonary disease
  * Active infections
  * Cancer (current or treated within the past 2 years) or coagulation disorder
  * Rapid weight change within the past year
  * Physically unable to participate in the intervention
  * Are currently taking, or recently (w/in 1 month of participation) taken prescribed, or over the counter ergogenic aids or compounds known to be banned by the NCAA.
  * Less than 16 years of age
  * Vegan patients
  * Patient over the age of 40
  * Pregnancy ( As part of standard of care, all female participants will be administered a urine pregnancy test prior to surgery. A negative test result is required to participate in the study.)
  * Any known or diagnosed kidney, GI, or liver disorders
  * Taking any medications known to affect protein metabolism. This includes, but is not limited to any drugs involved in hormone replacement therapy to treat conditions such as:

    * Hypothyroidism: example - levothyroxine
    * Hypogonadism: example - exogenous testosterone, estrogen, or any other forms of androgenic or anabolic hormone compounds
    * Growth hormone or growth hormone analogues
    * Type I or Type II diabetes requiring insulin
  * Currently taking protein supplements, amino acid supplements, or any known ergogenic aids.
  * Notably, all patients would need to confirm they will be doing their rehab through Houston Methodist
  * Patients diagnosed with protein intolerance or digestive issues associated with consuming protein

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | Pre-operation, 4, 8 and 12 weeks post-operation
  Lean mass in the effected limb

SECONDARY OUTCOMES:
Patient Reported Outcomes | Pre-operation 4, 8 and 12 weeks post-operation
  Knee injury and osteoarthritis outcome score (KOOS) JR Survey - This is a survey regarding pain and stiffness in the knee. Scales range from 1 (none) to 5 (extreme)
Patient Reported Outcomes | Pre-operation 4, 8 and 12 weeks post-operation
  Tampa Scale Survey - This is a patient perception scale of injury from a scale from 1 strongly disagree to 4 strongly agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No